CLINICAL TRIAL: NCT02537184
Title: Impact of Two Recall Intervals Associated to Oral Health Counseling on Dental Caries Incidence, Anxiety and Quality of Life of Preschool Children With High Caries Risk: Randomized Clinical Trial
Brief Title: Impact of Two Recall Intervals on Dental Caries Incidence and Other Outcomes of Preschool Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Thais Cordeschi, MSc student, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/17758-6
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2015-09-03 (Estimated); Status verified 2015-08

CONDITIONS: Dental Caries; Quality of Life; Anxiety
MeSH Terms: conditions — Dental Caries; Anxiety Disorders | interventions — Quality of Life; Time; Costs and Cost Analysis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - Recall Interval of 4 months (Other): Oral clinical conditions:
  Only at baseline all childrens will receive 5% sodium FV (Duraphat, Colgate Oral Pharmaceuticals). Caries incidence assessment dental anxiety assessment oral health related quality of life assessment time and costs assessment Procedure/Surgery: Oral clinical conditions Caries incidence assessment dental anxiety assessment oral health related quality of life assessment time and costs assessment
  Interventions: Procedure: Oral Clinical conditions
- Group 2 - Recall Interval of 8 months (Other): Oral clinical conditions:
  Only at baseline all childrens will receive 5% sodium FV (Duraphat, Colgate Oral Pharmaceuticals). Caries incidence assessment dental anxiety assessment oral health related quality of life assessment time and costs assessment Procedure/Surgery: Oral clinical conditions Caries incidence assessment dental anxiety assessment oral health related quality of life assessment time and costs assessment
  Interventions: Procedure: Oral Clinical conditions

INTERVENTIONS:
Procedure: Oral Clinical conditions — caries incidence assessment dental anxiety assessment
  Other Names: Caries Incidence; dental anxiety; oral health related quality of life; time and costs

SUMMARY:
Objectives: To assess the beneficial and harmful effects of two recall intervals on caries incidence (primary outcome) in preschool children with high caries risk. The level of anxiety, oral health related quality of life (OHRQoL), time and cost (secondary outcomes) according to each interval will also be assessed. Methods: The sample will consist of 224 children between 3-5 years of age, of both genders, with high caries risk according to the clinical criteria adapted from the Municipal Health Secretary of São Paulo. Children will be randomly allocated into two study groups: Group 1 (G1) - oral clinical examination + orientation for oral health and diet in return for 4 months; and Group 2 (G2) - oral clinical examination + orientation for oral health and diet in return for 8 months. An examiner calibrated and blinded to the study groups and the secondary outcomes will perform the clinical examinations, which consist of: gingival bleeding index, dental plaque index, detection of caries and its activity according to the ICDAS (International Caries Detection and Assessment System) and the clinical features of active and inactive caries lesions will be associated with the criteria discribed in ICDAS Commitee manual. An external dentist will conduct the assessment of the anxiety levels assessed by the Facial Image Scale, the OHRQoL measured by B-ECOHIS, the time and costs. All groups will be followed for an initial period of 16 months, totaling four follow-up visits for G1 and two follow-up visits to the G2. All analyzes will be performed by intention to treat (ITT) and considering the sensitivity analysis to assess the differences between the ITT analyzes and analyzes of complete cases.

DETAILED DESCRIPTION:
An examiner calibrated and blinded to the study groups and the secondary outcomes will perform the clinical examinations, which consist of: the gingival bleeding index, dental plaque index, detection of caries and its activity according to the ICDAS (International Caries Detection and Assessment System) and the clinical features of active and inactive caries lesions will be associated with the criteria discribed in ICDAS Commitee manual. An external dentist will conduct the assessment of the anxiety levels assessed by the Facial Image Scale, the OHRQoL measured by B-ECOHIS (Brazilian Early Childhood Oral Health Impact Scale), the time and costs. All groups will be followed for a period of 36 months. All analyzes will be performed with the intention of treatment (ITT) and considering the sensitivity analyzes to assess the differences between the ITT analyzes and the complete cases analyzes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* Children between 3-5 years of age, of both genders, with caries high risk according to the clinical criteria adapted from the Secretary of Health of São Paulo and enrolled in public schools.
* Guardians who have signed the informed consent confirming their participation and their child in research.

Exclusion Criteria:

* Children showing visible dental plaque and gingivitis in baseline.
* Children showing more than 06 active and/or inactive caries cavitated surfaces, and who show fistula and/or dental abscess.
* Special patients.
* Children who received professional application of fluoride in the 6 months prior to the

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 224 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Dental caries incidence | Baseline, 4 months and 8 months
  Dental caries will be assessed using the ICDAS criteria (Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, et al. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol 2007; 35: 170-8).

SECONDARY OUTCOMES:
Level of anxiety | Baseline, 4 months and 8 months
  Level of anxiety will be assessed using the Facial Image Scale (Buchanan H, Niven N. Validation of a facial image scale to assess child dental anxiety. Int J Paediatr Dent 2002;12:47-52)
Oral health related quality of life | Baseline, 4 months and 8 months
  Oral health related quality of life will be assessed using the Brazilian validation of the ECOHIS (Scarpelli AC, Oliveira BH, Tesch FC, Leão AT, Pordeus IA, Paiva SM. Psychometric properties of the Brazilian version of the Early Childhood Oral Health Impact Scale (B-ECOHIS). BMC Oral Health. 2011; 11:19).
Time | Baseline, 4 months and 8 months
  The time in minutes, used in the recall interval visits, will be recorded in four categories: time spent on clinical examination including prophylaxis, hygiene and diet orientations, and time spent when the patient miss the recall visit. The total time will correspond to the sum of these categories.
Costs | Baseline, 4 months and 8 months
  Costs in real (continuous variable) will be recorded in three categories: salary of the dentist and dental assistant paid in public dental services in São Paulo, cost of dental materials/products used in the appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Bonecker, Professor, Study Chair — University of Sao Paulo
Locations (1):
- Dental School of University of São Paulo, São Paulo, São Paulo, Brazil